CLINICAL TRIAL: NCT05608213
Title: Lenvatinib Plus Iodine-125 Seed Brachytherapy Compared With Lenvatinib Alone for TACE-refractory Hepatocellular Carcinoma: a Single Center, Prospective, Randomized Control Trail
Brief Title: Lenvatinib Plus I-125 Seed Brachytherapy vs. Lenvatinib for TACE-refractory HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-11
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Lenvatinib; iodion-125 seed
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Len-I (Experimental)
  Interventions: Procedure: Lenvatinib Plus I-125 Seed Brachytherapy
- Len (Active Comparator)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Procedure: Lenvatinib Plus I-125 Seed Brachytherapy — Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be administered to the patients. Iodion-125 seeds will be implanted into the the target lesions (viable intrahepatic tumor and/or vascular tumor thrombus) under CT guidance according to the pre-operative planning within 7 days after lenvatinib administration. Iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.
  Arms: Len-I
Drug: Lenvatinib — Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be administered to the patients.
  Arms: Len

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib plus iodine-125 seed brachytherapy (Len-I) compared with lenvatinib (Len) alone for patients with hepatocellular carcinoma (HCC) refractory to transarterial chemoembolization (TACE).

DETAILED DESCRIPTION:
This is a single-center, prospective and randomized controlled trial to evaluate the efficacy and safety of Len-I versus Len alone for patients with TACE-refractory HCC.

187 patients with TACE-refractory HCC will be enrolled in this study. The patients will receive either Len-I or Len alone using an 2:1 randomization scheme.

Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be administered to the patients and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. For patients in the Len-I arm, iodion-125 seeds will be implanted into the the target lesions (viable intrahepatic tumor and/or vascular tumor thrombus) under CT guidance according to the pre-operative planning within 7 days after lenvatinib administration. Iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.

The primary end point of this study is overall survival (OS). The secondary endpoints are progression-free survival (PFS), time to progression (TTP), objective response rate (ORR), disease control rate (DCR), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* HCC confirmed by histopathology and/or cytology, or diagnosed clinically
* Diagnosis of HCC with TACE refractoriness according to the criteria proposed by Japan Society of Hepatology (2021)
* Patients who have Tumor recurrence after surgical resection or ablation are allowed to be included
* At least one measurable intrahepatic target lesion
* Child-Pugh class A/B
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months

Exclusion Criteria:

* Extrahepatic metastasis
* Tumor thrombus involving main portal vein or both the first left and right branch of portal vein
* Vena cava invasion
* Patients who received prior systemic therapy, immunotherapy, hepatic arterial infusion chemotherapy (HAIC) or radiotherapy for HCC
* History of organ and cell transplantation
* History of bleeding from esophagogastric varices
* History of hepatic encephalopathy
* Hematologic examination: platelets <50×10^9/L
* Prothrombin time prolongation ≥ 4s
* Severe organ (heart, lung, kidney) dysfunction
* History of malignancy other than HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 4 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Time to Progression (TTP) | 4 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST).
Objective response rate (ORR) | 4 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
Disease control rate (DCR) | 4 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
Adverse Events (AEs) | 4 years
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China